CLINICAL TRIAL: NCT03934099
Title: A Randomized, Multicenter, Double-blind, Double-dummy, Parallel-group, Placebo and Active Comparator-controlled, Dose Finding, and Phase II Study to Assess Efficacy and Safety of LC350189 in Gout Patients With Hyperuricemia
Brief Title: A Study to Assess Efficay and Safety of LC350189 Different Doses in Gout Patients With Hyperuricemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-GDCL002
Record Dates: First submitted 2019-04-25; First posted 2019-05-01 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- LC350189 50mg (Experimental): LC350189 50mg, Once a day (QD)
  Interventions: Drug: LC350189 formulated capsule
- LC350189 100mg (Experimental): LC350189 100mg, QD
  Interventions: Drug: LC350189 formulated capsule
- LC350189 200mg (Experimental): LC350189 200mg, QD
  Interventions: Drug: LC350189 formulated capsule
- Placebo (Placebo Comparator): Placebo, QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LC350189 formulated capsule — Xanthine Oxidase Inhibitor
  Arms: LC350189 100mg; LC350189 200mg; LC350189 50mg
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The aim of this 12-week randomized multicenter double-blind parallel group placebo-controlled dose finding study is to assess the efficacy and safety of three different doses of LC350189 in subjects with hyperuricemia and a diagnosis of gout.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects or the subject's legally acceptable representatives who sign a written informed consent form prior to the initiation of any study procedures.
2. Subjects with hyperuricemia and a history or presence of gout per American College of Rheumatology (ACR) criteria.

Exclusion Criteria:

1. Subjects with secondary hyperuricemia (e.g., due to myeloproliferative disorder, or organ transplant).
2. Subjects experiencing an active acute gout attack within 3 weeks prior to screening (Visit 1).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyungjin Cho, MD, Study Director — LG Chem, Ltd.
Locations (33):
- United States (33):
  - Synexus Clinical Research, Birmingham, Alabama
  - Synexus Clinical Research, Chandler, Arizona
  - Synexus Clinical Research, Mesa, Arizona
  - Synexus Clinical Research, Tucson, Arizona
  - Preferred Research Partner, Little Rock, Arkansas
  - Health Awareness Inc, Jupiter, Florida
  - Meridien Research, Maitland, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Meridien Research, St. Petersburg, Florida
  - Clinical Research Trials of Florida, Inc, Tampa, Florida
  - Avita Clinical Trials, Tampa, Florida
  - IACT Health, Columbus, Georgia
  - Synexus Clinical Research, Chicago, Illinois
  - Synexus Clinical Research, Richfield, Minnesota
  - Olive Branch Family Medical Cente, Olive Branch, Mississippi
  - Synexus Clinical Research, St Louis, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Synexus Clinical Research, Omaha, Nebraska
  - Synexus Clinical Research, Henderson, Nevada
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Synexus Clinical Research, Akron, Ohio
  - Synexus Clinical Research, Cincinnati, Ohio
  - Synexus Clinical Research, Columbus, Ohio
  - Paramount Medical Research and Consulting, Middleburg Heights, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Synexus Clinical Research, Anderson, South Carolina
  - Avant Research Associates, Austin, Texas
  - Synexus Clinical Research, Dallas, Texas
  - Discovery MM Services Incorporated, Houston, Texas
  - Synexus Clinical Research, San Antonio, Texas
  - Synexus Clinical Research, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Dominion Medical Associates, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 156 participants enrolled, 13 were initially assigned to an active control group (Febuxostat) under the original protocol. This group was removed following a protocol amendment. Final results are reported based on the amended protocol, which excluded the active control group. Therefore, the discrepancy between the total number randomized and the final reported number reflects this change.
Period: Overall Study
Arm/Group | LC350189 50mg | LC350189 100mg | LC350189 200mg | Placebo
Started | 34 | 38 | 37 | 34
Completed | 30 | 32 | 34 | 32
Not Completed | 4 | 6 | 3 | 2
Not completed — Adverse Event | 0 | 3 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 1
Not completed — Other reasons | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LC350189 50mg | LC350189 100mg | LC350189 200mg | Placebo | Total
Number analyzed (Participants) | 34 | 38 | 37 | 34 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (9.60) | 56.6 (10.64) | 54.6 (10.66) | 55.4 (9.97) | 54.7 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 5 | 9
  Male | 33 | 37 | 35 | 29 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 7 | 7 | 30
  Not Hispanic or Latino | 28 | 28 | 30 | 27 | 113
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 2 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 0 | 3
  Black or African American | 3 | 6 | 6 | 5 | 20
  White | 30 | 27 | 25 | 29 | 111
  More than one race | 0 | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With sUA (Serum Uric Acid) < 5.0 mg/dL at Day 84
Description: sUA level was measured at Day 84
Time Frame: Day 84
Measure: Number; unit: Percentage of participants
Arm/Group | LC350189 50mg | LC350189 100mg | LC350189 200mg | Placebo
Number analyzed (Participants) | 34 | 38 | 37 | 34
Percentage of participants | 47.1 | 44.7 | 62.2 | 2.9

2. Secondary Outcome: Percentage of Participants With sUA (Serum Uric Acid) < 6.0 mg/dL at Day 84
Description: sUA level was measured at Day 84
Time Frame: Day 84
Measure: Number; unit: Percentage of participants
Arm/Group | LC350189 50mg | LC350189 100mg | LC350189 200mg | Placebo
Number analyzed (Participants) | 34 | 38 | 37 | 34
Percentage of participants | 58.8 | 63.2 | 78.4 | 2.9

3. Secondary Outcome: Maximum Percent Reduction in sUA (Serum Uric Acid) Level
Description: sUA level was measured at Day 1, 14, 28, 56, and 84
Time Frame: Up to Day 84
Measure: Mean (Standard Deviation); unit: Percentage of reduction in sUA
Arm/Group | LC350189 50mg | LC350189 100mg | LC350189 200mg | Placebo
Number analyzed (Participants) | 34 | 38 | 37 | 34
Percentage of reduction in sUA | -46.67 (13.560) | -50.64 (19.127) | -66.79 (15.787) | -11.20 (8.814)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | LC350189 50mg | LC350189 100mg | LC350189 200mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/38 | 0/37 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/38 | 0/37 | 0/34
Other Adverse Events (participants affected / at risk) | 15/34 | 13/38 | 21/37 | 8/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LC350189 50mg (N=34) | LC350189 100mg (N=38) | LC350189 200mg (N=37) | Placebo (N=34)
Diarrehoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Gout flare (Metabolism and nutrition disorders) | 9 (16) | 6 (11) | 10 (15) | 6 (6)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Coronavirus test positive (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2) | 6 (6) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT03934099/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT03934099/SAP_001.pdf